CLINICAL TRIAL: NCT03034902
Title: Detection of Area of Ischemia in Patients With Subacute Stroke Via a Hybrid EEG-fNIRS Brain-computer Interface
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The collaborating investigator has moved and cannot collect further data.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Paulina Sergot, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HSC-MS-16-0481
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Combined EEG and fNIRS (Experimental): EEG is electroencephalography. fNIRS is functional near infrared spectroscopy. The EEG+NIRS recordings will be obtained via an extended EEG cap that is applied to the subject's head. Changes in neuronal activity and hemodynamics will be measured.
  Interventions: Device: Combined EEG and fNIRS

INTERVENTIONS:
Device: Combined EEG and fNIRS — The EEG+NIRS recordings will be obtained via an extended EEG cap that is applied to the subject's head. Changes in neuronal activity and hemodynamics will be measured. The EEG component is the microEEG by BioSignal Group, UA. The fNIRS component is the NIRScout 24x32, NIRx Medizintechnik GmbH, Germany

SUMMARY:
The purpose of this research study is to determine whether a combined electroencephalography (EEG) and functional near infrared spectroscopy (fNIRS) recording is able to detect changes in brain activity and blood flow after stroke.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a subacute ischemic stroke with symptom onset within 8 weeks
* Must have a measurable deficit on the National Institute of Health Stroke Scale (NIHSS)
* Able to give and sign informed consent

Exclusion Criteria:

* Aphasia
* Underlying dementia
* Any chronic neurological disorder
* Malignancy
* Non-ambulatory (ambulation with assistance will be included)
* Modified Rankin Score (mRS) > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal blood flow as assessed by fNIRS | immediately at the time of combined EEG and fNIRS for up to 60 minutes
  Abnormal blood flow is determined by comparing a part of the patient's brain not affected by stroke to a part of the patient's brain affected by stroke.
Number of participants with abnormal neuronal activity as assessed by EEG | immediately at the time of combined EEG and fNIRS for up to 60 minutes
  Abnormal neuronal activity is determined by comparing a part of the patient's brain not affected by stroke to a part of the patient's brain affected by stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina B Sergot, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States